CLINICAL TRIAL: NCT04388384
Title: Neratinib in Patients With HER2+ Breast Cancer: a Multi-centric, Multi-national, Prospective, Longitudinal, Non-interventional Study in Germany, Austria and Switzerland
Brief Title: Real-life Pan-HER-blockade With Neratinib
Acronym: ELEANOR
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Pharma GmbH (Industry)
Collaborators: iOMEDICO AG (Industry); Pierre Fabre Pharma Austria (Unknown); Pierre Fabre Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS07075
Record Dates: First submitted 2020-05-05; First posted 2020-05-14 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2024-10

CONDITIONS: Breast Neoplasm
MeSH Terms: conditions — Breast Neoplasms | interventions — neratinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Neratinib — Neratinib standard dose 240 mg once daily for 1 year
  Other Names: Nerlynx

SUMMARY:
So far, there is no data available on treatment of patients with early-stage hormone receptor (HR) positive, human epidermal growth factor receptor 2 (HER2)-overexpressed/amplified breast cancer, who completed adjuvant trastuzumab-based therapy less than one year ago, in the clinical routine setting.

ELEANOR - designed as a prospective, longitudinal, non-interventional study (NIS) - will investigate real-world use of neratinib and its treatment management in patients with HR-positive, HER2-overexpressing/amplified breast cancer stage I-III having completed adjuvant trastuzumab-based therapy less than one year ago. Data from this study will contribute to a deeper understanding and characterization of the everyday use of neratinib in a broader patient population in the German and Austrian routine setting.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of the patient with regard to the pseudonymized documentation;
* Legally capable female patient ≥ 18 years of age (no upper limit);
* Decision was taken to treat the patient with neratinib in accordance with the current SmPC and by prescription; this decision was taken prior to and independent from the inclusion into the study;
* Treatment with neratinib is planned to be started;
* Hormone receptor (HR) positive, Human epidermal growth factor receptor 2 (HER2) overexpressing/amplified breast cancer stage I-III;
* Completion of prior trastuzumab-based therapy less than 1 year ago;
* No signs of relapse before initiation of neratinib treatment.

Exclusion Criteria:

* Presence of any contraindication with regard to the neratinib treatment as specified in the corresponding Summary of Product Characteristics (SmPC);
* Current or upcoming participation in an interventional clinical trial;
* Prisoners or persons who are compulsorily detained (involuntarily incarcerated)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female patients with HR-positive, HER2-overexpressing/amplified breast cancer stage I-III having completed adjuvant trastuzumab-based therapy less than one year ago and with a decision to receive extended adjuvant treatment with neratinib according to the current SmPC.
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Patient Compliance | 12 months of treatment
  Rate of patients being compliant to therapy with neratinib. A patient is defined as being compliant, if she has taken the prescribed neratinib dose for at least 75% of the treatment days.

SECONDARY OUTCOMES:
Patient profile at baseline | Baseline
  % of patients with different demographic characteristics
Disease profiles at baseline | Baseline
  % of patients with different disease characteristics
Pretreatment characteristics at baseline | Baseline
  % of patients with different pretreatments
Reason for neratinib treatment | Baseline
  % of patients with different reason for treatment selection (efficacy, safety profile, quality of life, patients preference, physician's preference, comorbidities, other)
Neratinib treatment characteristics | 12 months of treatment
  Absolute and relative dose intensity
Neratinib treatment characteristics | 12 months of treatment
  % of patients with dose modification
Neratinib treatment characteristics | 12 months of treatment
  % of patients with different reasons for dose modification (toxicity, concomitant disease, patient's wish, treatment holiday, other)
Neratinib treatment characteristics | 12 months of treatment
  % of patients with different concomitant medications
Relapse of disease | through study completion; maximum follow-up 55 months
  % of patients with relapse of disease
Patient reported outcome - EQ-5D-5L | 12 months of treatment
  The EQ-5D-5L is a standardized instrument for use as a measure of general health status preferences. It measures 5 dimensions of health including mobility, self-care, pain/discomfort, anxiety, and general health via a horizontal visual analog scale. Applicable to a wide range of health conditions and treatments, it provides a simple descriptive profile and a single index value for health status.
Patient reported outcome - STIDAT | 12 months of treatment
  The Systemic Therapy Induced Diarrhea Assessment Tool (STIDAT) questionnaire is a validated, patient-reported assessment tool designed to accurately identify the presence of diarrhea and its severity using multiple bowel habit dimensions in patients with systemic therapy-induced diarrhea (STID) of multiple solid tumors who received systemic therapy with or without radiation.
Physicians' treatment satisfaction: 5 point scale | 12 months of treatment
  % of patients with different physician satisfaction scores (5 point scale from very dissatisfied to very satisfied)
Patients' treatment satisfaction: 5 point scale | 12 months of treatment
  % of patients with different patient satisfaction scores (5 point scale from very dissatisfied to very satisfied)
Safety and tolerability of treatment with neratinib | 12 months of treatment + 30 days of safety follow-up
  % of patients with adverse events overall
Safety and tolerability of treatment with neratinib | 12 months of treatment + 30 days of safety follow-up
  % of patients with adverse events by intensity
Safety and tolerability of treatment with neratinib | 12 months of treatment + 30 days of safety follow-up
  Time to onset of first adverse event
Safety and tolerability of treatment with neratinib | 12 months of treatment + 30 days of safety follow-up
  Duration of adverse events
Safety and tolerability of treatment with neratinib | 12 months of treatment + 30 days of safety follow-up
  % of patients with action taken against adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Vannier, Dr, Study Director — Pierre Fabre Pharma GmbH
Locations (94):
- Austria (6):
  - Clinic, Klagenfurt, Carinthia
  - Clinic, Salzburg, Salzburg
  - Clinic, Schwarzach im Pongau, Salzburg
  - Clinic, Graz, Styria
  - Clinic, Vöcklabruck, Upper Austria
  - Clinic, Vienna, Vienna
- Germany (82):
  - Clinic, Baden-Baden, Baden-Wurttemberg
  - Community Health Center, Freiburg im Breisgau, Baden-Wurttemberg
  - Medical Practice, Heidelberg, Baden-Wurttemberg
  - Medical Practice, Heidenheim, Baden-Wurttemberg
  - Clinic, Nürtingen, Baden-Wurttemberg
  - Oncology Center, Offenburg, Baden-Wurttemberg
  - Clinic, Schwäbisch Hall, Baden-Wurttemberg
  - Medical Practice, Villingen-Schwenningen, Baden-Wurttemberg
  - Clinic, Weinheim, Baden-Wurttemberg
  - Clinic, Winnenden, Baden-Wurttemberg
  - Clinic, Ansbach, Bavaria
  - Medical Practice, Aschaffenburg, Bavaria
  - Practice, Augsburg, Bavaria
  - Clinic, Bamberg, Bavaria
  - Clinic, Deggendorf, Bavaria
  - Community Health Center, Eggenfelden, Bavaria
  - Clinic, Landshut, Bavaria
  - Community Health Center, Landshut, Bavaria
  - Clinic, Marktredwitz, Bavaria
  - Community Health Center, München, Bavaria
  - Clinic, München, Bavaria
  - Medical Practice, Bad Liebenwerda, Brandenburg
  - Clinic, Neuruppin, Brandenburg
  - Clinic, Potsdam, Brandenburg
  - Medical Practice, Bremen, City state Bremen
  - Clinic, Bremen, City state Bremen
  - Oncology Center, Hamburg, Hamburg
  - Clinic, Darmstadt, Hesse
  - Clinic, Frankfurt am Main, Hesse
  - Clinic, Wiesbaden, Hesse
  - Medical Care Center, Georgsmarienhütte, Lower Saxony
  - Community Health Center, Goslar, Lower Saxony
  - Practice, Göttingen, Lower Saxony
  - Clinic, Hanover, Lower Saxony
  - Medical Practice, Hildesheim, Lower Saxony
  - Medical Practice, Leer, Lower Saxony
  - Clinic, Lüneburg, Lower Saxony
  - Clinic, Oldenburg, Lower Saxony
  - Medical Practice, Uelzen, Lower Saxony
  - Medical Practice, Westerstede, Lower Saxony
  - Medical Practice, Wilhelmshaven, Lower Saxony
  - Medical Practice, Greifswald, Meckelnburg-Vorpommern
  - Clinic, Rostock, Mecklenburg-Vorpommern
  - Medical Practice, Stralsund, Mecklenburg-Vorpommern
  - Medical Practice, Bonn, North Rhine-Westphalia
  - Medical Practice, Bottrop, North Rhine-Westphalia
  - Clinic, Cologne, North Rhine-Westphalia
  - Clinic, Datteln, North Rhine-Westphalia
  - Clininc, Essen, North Rhine-Westphalia
  - Medical Practice, Gütersloh, North Rhine-Westphalia
  - Clinic, Hamm, North Rhine-Westphalia
  - Medical Practice, Moers, North Rhine-Westphalia
  - Medical Practice, Mülheim, North Rhine-Westphalia
  - Community Health Center, Neuss, North Rhine-Westphalia
  - Community Health Center, Soest, North Rhine-Westphalia
  - Medical Practice, Troisdorf, North Rhine-Westphalia
  - Clinic, Witten, North Rhine-Westphalia
  - Medical Practice, Mayen, Rhineland-Palatinate
  - Clinic, Neustadt, Rhineland-Palatinate
  - Clinic, Chemnitz, Saxony
  - Oncology Center, Dresden, Saxony
  - Medical Praxis, Freital, Saxony
  - Clinic, Leipzig, Saxony
  - Medical Practice, Plauen, Saxony
  - Medical Practice, Burg, Saxony-Anhalt
  - Medical Practice, Halle, Saxony-Anhalt
  - Clinic, Magdeburg, Saxony-Anhalt
  - Clinic, Quedlinburg, Saxony-Anhalt
  - Clinic, Salzwedel, Saxony-Anhalt
  - Clinic, Stendal, Saxony-Anhalt
  - Clinic, Eutin, Schleswig-Holstein
  - Medical Practice, Berlin, State of Berlin
  - Clinical Practice, Berlin, State of Berlin
  - Medical Care center, Neuwied, Theinland-Pfalz
  - Medical Practice, Erfurt, Thuringia
  - Medical Practice, Hildburghausen, Thuringia
  - Clinic, Jena, Thuringia
  - Medical Practice, Meiningen, Thuringia
  - Oncology Center, Neuhaus am Rennweg, Thuringia
  - Medical Care Center, Saalfeld, Thuringia
  - Clinic, Suhl, Thuringia
  - Medical Practice, Suhl, Thuringia
- Switzerland (6):
  - Practice, Basel, Canton of Basel-City
  - Practice, Biel/Bienne, Canton of Bern
  - Clinic, Olten, Canton of Solothurn
  - Clinic, Lausanne, Canton of Vaud
  - Clinic, Zurich, Canton of Zurich
  - Clinic, Chur, Kanton Graubünden

IPD SHARING:
Plan to Share IPD: No